CLINICAL TRIAL: NCT05333198
Title: Effects of Oculomotor and Vestibular Ocular Reflex Exercises on Vertigo, Dizziness and Balance in Patients With Benign Paroxysmal Positional Vertigo
Brief Title: Oculomotor and Vestibular Ocular Reflex Exercises in Patients With Benign Paroxysmal Positional Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Ezza Zikrea
Record Dates: First submitted 2022-01-21; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Benign Paroxysmal Positional Vertigo (Disorder)
Keywords: Benign Paroxysmal Positional Vertigo; Oculomotor exercises; Vestibular Ocular Reflex (VOR) exercises
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Motor Activity | interventions — Reflex, Vestibulo-Ocular; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy using Epley's maneuver (Other): Epley's maneuver was performed once a week for three weeks. The maneuver was performed by patient in sitting position, head was rotated towards involved side and then extended to 30 degrees, it was then rotated to 180 degrees followed by patient rolling onto opposite side. Each position was maintained for 1-2 minutes.
  Interventions: Other: Traditional physical therapy using Epley's maneuver
- Oculomotor and Vestibular Ocular Reflex (VOR) exercises (Active Comparator): oculomotor and VOR exercises after Epley's maneuver. The exercises were performed for approximately 5 minutes daily or 1 to 2 minutes, 3 to 4 times a day, in sitting position. The exercises were continued for three weeks. The maneuver was performed by patient in sitting position, head was rotated towards involved side and then extended to 30 degrees, it was then rotated to 180 degrees followed by patient rolling onto opposite side. Each position was maintained for 1-2 minutes. Saccadic exercises were performed by moving eyes between two stationary targets. Smooth pursuit exercises were performed by tracking a moving target while keeping head still and VOR exercises were performed by moving head left to right while maintaining eyes on stationary target
  Interventions: Other: Oculomotor and Vestibular Ocular Reflex (VOR) exercises

INTERVENTIONS:
Other: Traditional physical therapy using Epley's maneuver — Epley's maneuver was performed once a week for three weeks. The maneuver was performed by patient in sitting position, head was rotated towards involved side and then extended to 30 degrees, it was then rotated to 180 degrees followed by patient rolling onto opposite side. Each position was maintained for 1-2 minutes.
  Arms: Traditional physical therapy using Epley's maneuver
Other: Oculomotor and Vestibular Ocular Reflex (VOR) exercises — oculomotor and VOR exercises after Epley's maneuver. The exercises were performed for approximately 5 minutes daily or 1 to 2 minutes, 3 to 4 times a day, in sitting position. The exercises were continued for three weeks. The maneuver was performed by patient in sitting position, head was rotated towards involved side and then extended to 30 degrees, it was then rotated to 180 degrees followed by patient rolling onto opposite side. Each position was maintained for 1-2 minutes. Saccadic exercises were performed by moving eyes between two stationary targets. Smooth pursuit exercises were performed by tracking a moving target while keeping head still and VOR exercises were performed by moving head left to right while maintaining eyes on stationary target
  Arms: Oculomotor and Vestibular Ocular Reflex (VOR) exercises

SUMMARY:
The aim of this research is to assess effects of Oculomotor and VOR exercises on vertigo, dizziness and balance in patients with BPPV. Randomized controlled trial was conducted at Hameed Latif Hospital, Lahore. The sample size 32 participants which were divided into two groups, 16 participants in traditional physical therapy group and 16 in oculomotor and vestibular ocular reflex exercises group. Study duration was of 6 months. Sampling technique applied was non-probability consecutive sampling technique. Only 30-70 years individuals with Benign Paroxysmal Positional Vertigo (BPPV) were included. Tools used in the study are vertigo handicap questionnaire, visual vertigo analogue scale, dizziness handicap inventory, berg balance scale and dynamic gait index. The data was analyzed using SPSS.

DETAILED DESCRIPTION:
Randomized controlled trial was conducted at Hameed Latif Hospital, Lahore. The sample size 32 participants which were divided into two groups, 16 participants in traditional physical therapy group and 16 in oculomotor and vestibular ocular reflex exercises group. Study duration was of 6 months. Sampling technique applied was non-probability consecutive sampling technique. Only 30-70 years individuals with Benign Paroxysmal Positional Vertigo (BPPV) were included. Tools used in the study are vertigo handicap questionnaire, visual vertigo analogue scale, dizziness handicap inventory, berg balance scale and dynamic gait index. The data was analyzed using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have vertigo with posterior canal involvement during Dix-Hallpike test with or without accompanying nystagmus (objective or subjective BPPV).
* Ability to walk at least 3 meters by itself with or without assistive device
* Normal vision with or without correction by spectacles or contact lenses

Exclusion Criteria:

* Patients with other neurologic conditions, orthopedic problems, and uncontrolled metabolic diseases to eliminate confounding factors affecting balance performance
* Unable to understand and answer a simple verbal command.
* Previously underwent oculomotor and vestibular ocular exercises.
* Other vestibular disorders like Meniere disease
* Long-term use of benzodiazepines (more than 20 years).
* Patients who are already performing structured physical activities such as muscle strengthening exercises, Pilates, yoga or high intensity aerobic exercises

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Vertigo Handicap Questionnaire | First reading at 0 day
  It assess effect of vertigo on disability, handicap and benefits following therapeutic intervention both physically and psychologically.
Vertigo Handicap Questionnaire | second reading after 3 weeks
  It assess effect of vertigo on disability, handicap and benefits following therapeutic intervention both physically and psychologically.
Visual Vertigo Analogue Scale | First reading at 0 day
  Intensity of visual vertigo in nine challenging situations of visual motions that typically provoke dizziness
Visual Vertigo Analogue Scale | second reading after 3 weeks
  Intensity of visual vertigo in nine challenging situations of visual motions that typically provoke dizziness
Dizziness Handicap Inventory | First reading at 0 day
  Self-perceived handicapping effects imposed by dizziness.
Dizziness Handicap Inventory | second reading after 3 weeks
  Self-perceived handicapping effects imposed by dizziness.
Berg Balance Scale | First reading at 0 day
  Objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks
Berg Balance Scale | First reading at 3 week
  Objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks
Dynamic Gait Index | first reading after 0 day
  The clinical tool to assess gait, balance and fall risk. It evaluates not only usual steady-state walking, but also walking during more challenging tasks.
Dynamic Gait Index | second reading after 3 weeks
  The clinical tool to assess gait, balance and fall risk. It evaluates not only usual steady-state walking, but also walking during more challenging tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Binash Afzal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim HJ, Lee JO, Choi JY, Kim JS. Etiologic distribution of dizziness and vertigo in a referral-based dizziness clinic in South Korea. J Neurol. 2020 Aug;267(8):2252-2259. doi: 10.1007/s00415-020-09831-2. Epub 2020 Apr 16. PMID 32300888
- [Background] Scocco DH, Garcia IE, Barreiro MA. Sitting Up Vertigo. Proposed Variant of Posterior Canal Benign Paroxysmal Positional Vertigo. Otol Neurotol. 2019 Apr;40(4):497-503. doi: 10.1097/MAO.0000000000002157. PMID 30870365
- [Background] Dunlap PM, Holmberg JM, Whitney SL. Vestibular rehabilitation: advances in peripheral and central vestibular disorders. Curr Opin Neurol. 2019 Feb;32(1):137-144. doi: 10.1097/WCO.0000000000000632. PMID 30461465
- [Background] Wu P, Cao W, Hu Y, Li H. Effects of vestibular rehabilitation, with or without betahistine, on managing residual dizziness after successful repositioning manoeuvres in patients with benign paroxysmal positional vertigo: a protocol for a randomised controlled trial. BMJ Open. 2019 Jun 18;9(6):e026711. doi: 10.1136/bmjopen-2018-026711. PMID 31217316
- [Background] Kane AW, Diaz DS, Moore C. Physical Therapy Management of Adults with Mild Traumatic Brain Injury. Semin Speech Lang. 2019 Feb;40(1):36-47. doi: 10.1055/s-0038-1676652. Epub 2019 Jan 7. PMID 30616293
- [Background] Hillier S, McDonnell M. Is vestibular rehabilitation effective in improving dizziness and function after unilateral peripheral vestibular hypofunction? An abridged version of a Cochrane Review. Eur J Phys Rehabil Med. 2016 Aug;52(4):541-56. Epub 2016 Jul 12. PMID 27406654
- [Background] Arnold SA, Stewart AM, Moor HM, Karl RC, Reneker JC. The Effectiveness of Vestibular Rehabilitation Interventions in Treating Unilateral Peripheral Vestibular Disorders: A Systematic Review. Physiother Res Int. 2017 Jul;22(3). doi: 10.1002/pri.1635. Epub 2015 Jun 25. PMID 26111348
- [Background] Meldrum D, Burrows L, Cakrt O, Kerkeni H, Lopez C, Tjernstrom F, Vereeck L, Zur O, Jahn K. Vestibular rehabilitation in Europe: a survey of clinical and research practice. J Neurol. 2020 Dec;267(Suppl 1):24-35. doi: 10.1007/s00415-020-10228-4. Epub 2020 Oct 13. PMID 33048219
- [Background] Mempouo E, Lau K, Green F, Bowes C, Ray J. Customised vestibular rehabilitation with the addition of virtual reality based therapy in the management of persistent postural-perceptual dizziness. J Laryngol Otol. 2021 Oct;135(10):887-891. doi: 10.1017/S0022215121002127. Epub 2021 Aug 10. PMID 34372958
- [Background] Lin SI, Tsai YJ, Lee PY. Balance performance when responding to visual stimuli in patients with Benign Paroxysmal Positional Vertigo (BPPV). J Vestib Res. 2020;30(4):267-274. doi: 10.3233/VES-200709. PMID 32925126